CLINICAL TRIAL: NCT02996175
Title: Treatment of Sleep Disturbances in School-age Children With Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R21HD082307-01A1 (NIH)
Record Dates: First submitted 2015-11-30; First posted 2016-12-19 (Estimated); Last update posted 2018-06-04 (Actual); Status verified 2018-06

CONDITIONS: Down Syndrome
Keywords: Behavior; Sleep; Problems; Intervention
MeSH Terms: conditions — Down Syndrome; Behavior

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SMART (Experimental): Treatment group targeting behavioral sleep problems for 5 weeks.
  1. Introduction to the treatment program, an overview of common sleep problems in DS, and the basic principles of the behavioral approach as it relates to sleep problems
  2. Information on healthy sleep hygiene, preventative techniques, and use of visual supports
  3. Information on reinforcement and extinction procedures for bedtime struggles, codependence, night waking, early waking
  4. Information on procedures for delayed sleep onset and problematic sleep associations
  5. Feedback on implementation of behavioral sleep treatments and strategies for managing sleep hygiene in the future
  Interventions: Behavioral: Behavioral Sleep Treatment
- WISE (Active Comparator): Standard of care sleep treatment enhanced with psychoeducation. 1 Introduction to the general-education program, build rapport with family, and review basic information on Down syndrome 2 Introduction to understanding and interpreting results from clinical evaluations 3 Introduction to educational planning, expectations, and transition planning 4 Introduction to lifespan development and advocacy and support services available 5 Feedback on current concerns and methods for obtaining services to manage concerns
  Interventions: Behavioral: Standard of care sleep treatment enhanced with psychoeducation

INTERVENTIONS:
Behavioral: Behavioral Sleep Treatment — 1. Introduction to the treatment program, an overview of common sleep problems in DS, and the basic principles of the behavioral approach as it relates to sleep problems
  2. Information on healthy sleep hygiene, preventative techniques, and use of visual supports
  3. Information on reinforcement and extinction procedures for bedtime struggles, codependence, night waking, early waking
  4. Information on procedures for delayed sleep onset and problematic sleep associations
  5. Feedback on implementation of behavioral sleep treatments and strategies for managing sleep hygiene in the future
  Arms: SMART
Behavioral: Standard of care sleep treatment enhanced with psychoeducation — 1. Introduction to the general-education program, build rapport with family, and review basic information on Down syndrome
  2. Introduction to understanding and interpreting results from clinical evaluations
  3. Introduction to educational planning, expectations, and transition planning
  4. Introduction to lifespan development and advocacy and support services available
  5. Feedback on current concerns and methods for obtaining services to manage concerns
  Arms: WISE

SUMMARY:
The investigators long-term goal is to improve outcomes for children with Down syndrome (DS) and their caregivers. Towards that goal, the investigators propose a randomized clinical trial of a behavioral sleep treatment designed specifically for children with DS, documenting the impact not only on sleep, but also on the child's daytime inhibitory control and behavior problems, and the caregiver's sleep and stress levels. The investigators will randomize 80 families of children with DS ages 6-17 to receive either a 5-session behavioral sleep treatment (BST; targeting sleep education, behavioral principles and visual supports) or a general-education control condition (CON). The BST will cater to the unique needs of children with DS, adapting an intervention that successfully treats behavioral sleep disturbances in children with autism1. Pre- and post-intervention, children will undergo comprehensive assessments of cognitive, behavioral, and adaptive functioning involving direct testing and input from parents and teachers. Child and parent sleep will be monitored via actigraphy and parent-completed sleep diaries, and parents will report on their stress levels and mood.

DETAILED DESCRIPTION:
The investigators long-term goal is to improve outcomes for children with DS and their caregivers. Towards that goal, the investigators propose a randomized clinical trial of a behavioral sleep treatment designed specifically for children with DS, documenting the impact not only on sleep, but also on the child's daytime inhibitory control and behavior problems, and the caregiver's sleep and stress levels. The investigators will randomize 80 families of children with DS ages 6-17 to receive either a 5-session behavioral sleep treatment (BST; targeting sleep education, behavioral principles and visual supports) or a general-education control condition (CON). The BST will catered to the unique needs of children with DS, adapting an intervention developed by a member of the investigators research team with NIH support (R34 MH082882) that successfully treats behavioral sleep disturbances in children with autism41. Pre- and post-intervention, children will undergo comprehensive assessments of cognitive, behavioral, and adaptive functioning involving direct testing and input from parents and teachers. Child and parent sleep will be monitored via actigraphy and parent-completed sleep diaries, and parents will report on their stress levels and mood. As a critical first step towards an effective treatment, this initial efficacy study will address 3 aims:

Aim #1: Test the efficacy of manualized BST for improving the sleep of children with DS.

Hypothesis 1: Sleep duration and quality will improve more in the BST condition than the CON condition.

Aim #2: Test the impact of the BST on the daytime functioning of children with DS.

Hypothesis 2: Children receiving BST will make greater gains in inhibitory control, general behavior problems and other measures of executive dysfunction than in the CON condition.

Aim #3: Test whether the BST, which focuses on the child's sleep, also impacts caregivers' sleep and stress.

Hypothesis 3: Parents of children receiving BST will have improved sleep duration and decreased stress.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Down Syndrome
* 6-17 years of age
* behavioral sleep problem (presence of 5 or more nights a week of: bedtime resistance, delayed sleep onset, problematic sleep associations, nighttime awakenings or morning awakenings)
* English as primary language

Exclusion Criteria:

* past diagnosis of Pervasive Developmental Disorder-Not Otherwise Specified/Autism Spectrum Disorder
* History of blindness,deafness,motor impairment
* nonverbal mental age below 36 months
* any medication change w/in past 2 months affecting sleep

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2015-07; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Longer child sleep duration as measured by actigraphy and Improved sleep quality for child measure by Children's Sleep Habits Questionnaire (CSHQ) | Baseline, 6 Weeks, 19 Weeks
  33-item Parent reported sleep quality for Child over past week. Each item is scored 1-3 (1 = Rarely, 0-1x/week; 2 = Sometimes, 2-4x/week; 3= Usually, 5-7x/week). There are 6 questions with reverse scoring. This will yield a total between 33 and 99.
  This will be acquired from parent three times throughout study, data scored and entered into SPSS by coordinator using total score data for comparatives to actigraph results for total sleep.

SECONDARY OUTCOMES:
Improved child behaviors as measured by parent report on Child Behavior Checklist (CBCL) | Baseline, 6 Weeks, 19 Weeks
  113-Item parent report measure for child behavior now. Each item is scored 0-2 (0 = Not True (as far as you know); 1 = Somewhat or Sometimes True; 2 = Very True or Often True. Scoring is done through software giving T-scores for 8 subscales with borderline and clinical ranges identified. SPSS will be used for analysis to compare to parent report data from a daily behavior journal.
Longer Parent sleep duration as measured by actigraphy and reduced parental stress as measured by the Family Impact Questionnaire (FIQ). | Baseline, 6 Weeks, 19 Weeks
  50-item parent report measure rating child's impact on family and different areas of family functioning. Each of the first 48 items are scored 1-4 (1 = Not at all; 2 = Somewhat; 3 = Much; 4 = Very Much) and items 48 & 49 scored 1-7 (1 = Much Easier; 2 = Easier; 3 = Slightly Easier; 4 = About the Same; 5 = Slightly More Difficult; 6 = More Difficult; 7 = Much More Difficult). There are 5 items that are reverse scored. Scoring yields T-scores for 7 subscales.Data will be entered into SPSS and used as a parental stress scale for social impact.

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States